CLINICAL TRIAL: NCT01632826
Title: A Multicenter, Single-Arm, Open-Label Treatment Use Protocol for Pomalidomide (POM) in Combination With Low Dose Dexamethasone (LD-Dex) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Pomalidomide (POM) in Combination With Low Dose Dexamethasone (LD-Dex) in Patients With Relapsed or Refractory Multiple Myeloma
Acronym: PEXIUS
Status: Approved for marketing | Type: Expanded Access
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-4047-MM-009
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; refractory multiple myeloma; pomalidomide
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — 4 mg daily for 21 days in a 28 day cycle until disease progression or other reasons for treatment discontinuation

SUMMARY:
To provide pomalidomide access to relapsed/refractory multiple myeloma subjects with a likelihood of benefit from the pomalidomide treatment while the medication is not commercially available

DETAILED DESCRIPTION:
Several clinical studies indicate that pomalidomide has activity in relapsed and refractory multiple myeloma with response rates ranging between 30% and 60% at pomalidomide doses at 2 mg/day and/or 4 mg/day.

ELIGIBILITY:
Inclusion Criteria:

1. Must have documented diagnosis of relapsed or relapsed/refractory multiple myeloma and have measurable disease (serum or urine M-protein)
2. Age ≥ 18 years
3. Must have had at least ≥ 2 prior anti-myeloma therapies
4. Must have received at least 2 consecutive cycles of both lenalidomide and bortezomib, either alone or in combination
5. Must have failed treatment with the last lenalidomide-containing regimen and the last bortezomib-containing regimen
6. Must have documented disease progression during or after the last antimyeloma regimen
7. Females of childbearing potential (FCBP) must agree to utilize two reliable forms of contraception simultaneously or practice complete abstinence from heterosexual contact for at least 28 days before starting drug, while participating in the study and for at least 28 days after study treatment discontinuation.
8. Males must agree to use a latex condom during sexual contact with FCBP while participating in the study and for 28 days following discontinuation from study treatment.

Exclusion Criteria:

1. Peripheral Neuropathy ≥ Grade 2
2. Non-secretory multiple myeloma
3. Previous therapy with pomalidomide
4. Use of any investigational agents within 28 days or 5 half lives (whichever is longer) of initiating study treatment
5. Subjects with conditions requiring chronic steroid or immunosuppressive treatment.
6. Hypersensitivity to thalidomide, lenalidomide or dexamethasone
7. Known Human Immunodeficiency Virus positive, active or chronic Hepatitis A, B or C
8. Pregnant or breastfeeding females
9. Unacceptable hematological or biochemical laboratory abnormalities

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lars Sternas, MD, PhD, Study Director — Celgene Corporation
Locations (39):
- United States (24):
  - Celgene Study Site, Duarte, California
  - Celgene Study Site, Greenbrae, California
  - Celgene Study Site, Los Angeles, California
  - Celgene Study Site, Denver, Colorado
  - Celgene Study Site, West Palm Beach, Florida
  - Celgene Study Site, Marietta, Georgia
  - Celgene Study Site, Peoria, Illinois
  - Celgene Study Site, Indianapolis, Indiana
  - Celgene Study Site, Iowa City, Iowa
  - Celgene Study Site, Baltimore, Maryland
  - Celgene Study Site, Hyannis, Massachusetts
  - Celgene Study Site, St Louis, Missouri
  - Celgene Study Site, Omaha, Nebraska
  - Celgene Study Site, Hackensack, New Jersey
  - Celgene Study Site, New York, New York
  - Celgene Study Site, Philadelphia, Pennsylvania
  - Celgene Study Site, Sellersville, Pennsylvania
  - Celgene Study Site, Greenville, South Carolina
  - Celgene Study Site, Sioux Falls, South Dakota
  - Celgene Study Site, Dallas, Texas
  - Celgene Study Site, Houston, Texas
  - Celgene Study Site, Salt Lake City, Utah
  - Celgene Study Site, Morgantown, West Virginia
  - Celgene Study Site, Milwaukee, Wisconsin
- Canada (15):
  - Celgene Study Site, Calgary, Alberta
  - Celgene Study Site, Edmonton, Alberta
  - Celgene Study Site, Vancouver, British Columbia
  - Celgene Study Site, Victoria, British Columbia
  - Celgene Study Site, Winnipeg, Manitoba
  - Celgene Study Site, St. John's, Newfoundland and Labrador
  - Celgene Study Site, Halifax, Nova Scotia
  - Celgene Study Site, Hamilton, Ontario
  - Celgene Study Site, London, Ontario
  - Celgene Study Site, Ottawa, Ontario
  - Celgene Study Site, Toronto, Ontario
  - Celgene Study Site, Windsor, Ontario
  - Celgene Study Site, Montreal, Quebec
  - Celgene Study Site, Québec, Quebec
  - Celgene Study Site, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Qian X, Dimopoulos MA, Amatangelo M, Bjorklund C, Towfic F, Flynt E, Weisel KC, Ocio EM, Yu X, Peluso T, Sternas L, Zaki M, Moreau P, Thakurta A. Cereblon gene expression and correlation with clinical outcomes in patients with relapsed/refractory multiple myeloma treated with pomalidomide: an analysis of STRATUS. Leuk Lymphoma. 2019 Feb;60(2):462-470. doi: 10.1080/10428194.2018.1485915. Epub 2018 Aug 2. PMID 30068263